CLINICAL TRIAL: NCT07096375
Title: Competency of Coupling of IPACK Block With Adductor Canal Block Versus Adductor Canal Block Alone on Postoperative Pain, Functional Recovery and Inflammatory Response After Total Knee Replacement
Brief Title: Coupling of IPACK Block With Adductor Canal Block Versus Adductor Canal Block Alone on Pain, Functional Recovery and Inflammatory Response After Knee Replacement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD187/2024
Record Dates: First submitted 2025-06-15; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-11

CONDITIONS: Adductor Canal Block; Total Knee Replacement Surgery; Functional Recovery
Keywords: IPACK block; Adductor Canal Block; Inflammatory Response
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor canal block (ACB) + IPACK block (Active Comparator): Group A: 25 patients will receive adductor canal block under ultrasound using 20 ml bupivacaine 0.25% and IPACK block under direct visualization of ultrasound using 15 ml bupivacaine 0.25% at the start of surgery.
  IPACK Block which the patient will be placed in a supine position and knee will be placed in position of 90° flexion. A low-frequency ultrasound probe will be positioned in the popliteal crease, and a spinal needle will be inserted from the medial aspect of the knee from anteromedial to posterolateral direction in a plane between the popliteal artery and the femur. The tip of the needle will be placed 1-2 cm beyond the lateral edge of the artery, and 15 ml of bupivacaine 0.25% will be injected after negative aspiration.
  Interventions: Procedure: Adductor Canal Block (ACB) + iPACK Block
- Adductor Canal Block (ACB) + IPACK (sham injection) (Sham Comparator): Group B : 25 patients will receive Adductor canal block only under ultrasound guide using 20ml bupivacaine 0.25% and IPACK block under direct visualization of ultrasound using 15 ml of saline (sham injection) at the start of the surgery. The patients in Group B will receive ACB and IPACK block (sham injection) as described above.
  Interventions: Procedure: Adductor Canal Block (ACB) + iPACK Block (sham injection)

INTERVENTIONS:
Procedure: Adductor Canal Block (ACB) + iPACK Block — Adductor Canal Block (ACB) in the immediate preoperative period under a high-frequency ultrasound guidance in which the adductor canal is identified beneath the sartorius muscle and 20 ml of bupivacaine 0.25% will be injected in the canal using a 22-gaugusing a 22-gauge 100-mm short-bevelled regional block needle.
  IPACK Block which the patient will be placed in a supine position and knee will be placed in position of 90° flexion. A low-frequency ultrasound probe will be positioned in the popliteal crease, and a spinal needle will be inserted from the medial aspect of the knee from anteromedial to posterolateral direction in a plane between the popliteal artery and the femur. The tip of the needle will be placed 1-2 cm beyond the lateral edge of the artery, and 15 ml of bupivacaine 0.25% will be injected after negative aspiration.
  Other Names: Adductor Canal Block (ACB); IPACK block
  Arms: Adductor canal block (ACB) + IPACK block
Procedure: Adductor Canal Block (ACB) + iPACK Block (sham injection) — All patients will receive Adductor Canal Block in the immediate preoperative period under a high-frequency ultrasound guidance in which the adductor canal is identified beneath the sartorius muscle and 20 ml of bupivacaine 0.25% will be injected in the canal using a 22-gauge 100-mm short-bevelled regional block needle IPACK block which the patient will be placed in a supine position and knee will be placed in position of 90° flexion. A low-frequency ultrasound probe will be positioned in the popliteal crease, and a spinal needle will be inserted from the medial aspect of the knee from anteromedial to posterolateral direction in a plane between the popliteal artery and the femur. The tip of the needle will be placed 1-2 cm beyond the lateral edge of the artery, and 15 ml of normal saline will be injected after negative aspiration.
  Other Names: Adductor Canal Block; IPACK Block (sham injection)
  Arms: Adductor Canal Block (ACB) + IPACK (sham injection)

SUMMARY:
The aim of this study is to compare the Competency of coupling of IPACK Block with Adductor Canal Block versus Adductor Canal Block Alone on Postoperative Pain after total knee replacement as well as Functional Recovery and Inflammatory Response and range of motion postoperatively.

DETAILED DESCRIPTION:
Postoperative Analgesia Management and Evaluation of Outcomes:

After the total knee arthroplasty ended, the patients will be transmitted to the post anaesthesia care unit (PACU). The same multimodal postoperative analgesia will be applied in the PACU in three groups, which will be consistent with ketorolac 50 mg every twelve hours and acetaminophen 1 g i.v. every eight hours will be both applied for 3 days. If the NRS score is higher than 4, 5 mg morphine will be administered as rescue analgesia. Eight mg of odanesteron will be given when severe nausea or vomiting occurs. Enoxaparin for four weeks postoperatively will be given as a thromboembolism prophylaxis. Finally, patients will be ambulated with the help of the walker after the first ten postoperative hours.

Assessment of outcomes:

Primary outcome:

Assessment of pain after completing the surgical procedure and wear off of spinal analgesia that will be confirmed by Bromage scale and cold sensation.

The total cumulative dose of used morphine to control pain from the postoperative in post anaesthesia care unit and in orthopaedic wards. Also, total opioid consumption will be recorded at 0-6, 6-12, and 12-24 h after surgery as primary outcome of the study.

Secondary outcome:

The secondary outcomes including assessment of pain by visual analogue scale (VAS) will be done postoperatively at 8 hours, 12 hours and 24 hours postoperatively.

Visual analogue scale (VAS) (scale 0-10, where 0 = no pain and 10 = worst imaginable pain). All the patients will have the VAS score explained and taught for self-assessment of pain at the time of enrolment for the study (Bringuier et al., 2009).

As well as the range of motion and quadriceps strength will be measured to grade the functional recovery of the knee joint after surgery after the first ten hours postoperatively. The protractor will be used for the range of motion. The interval of activities will be recorded three times a day, 6 h apart, and i will use the best value as the day's value. The quadriceps strength will be measured by asking the patient to flex the hip and knee and the complete knee extension. The outcome assessor will use resistance to knee extension and palpated the thigh muscles to measure muscle strength. No muscle movement will score 0 points, no joint movement with muscle contraction will score 1 point, no gravity resistance with joint movement will score 2 points, gravity resistance will score 3 points, partial counterforce resistance with gravity resistance will score 4 points, and normal joint function will score 5 points.

Also, blood samples for neutrophil-lymphocytic ratio (NLR) and platelet-lymphocytic ratio (PLR) will be collected at 12 and 24 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee replacement.
* ASA physical status I to III
* Sex (males and females).
* Age 20 - 70 years.

Exclusion Criteria:

* Patients undergoing bilateral or revision total knee replacement.
* ASA physical status more than III
* Age less than 20 or older than 70
* severe renal insufficiency ( Estimated Glomerular filtration rate eGFR < 15 mL/min/1.73 m2 ).
* history of arrhythmia or seizures.
* Hypersensitivity to local anesthetics.
* Preexisting peripheral neuropathy and prior vascular surgery on femoral vessels on operated site.
* Infection near site of injection e.g. osteomyelitis, septic knee joint, etc.
* Patient refusal or with difficulties in comprehending numeric pain rating scale (NRS) pain scores
* Any contraindications for spinal anesthesia. (eg.: refusal of patients, coagulopathy, use of anticoagulants or antiplatelets...)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to compare the Competency of coupling of IPACK Block with Adductor Canal Block versus Adductor Canal Block Alone on Postoperative Pain after total knee replacement. | At 0 hour -6 hours, 6 hours-12 hours and 12 hours - 24 hours after surgery
  Total cumulative dose of used morphine (mg) to control pain will be recorded at 0 hour -6 hours, 6 hours -12 hours and 12 hours - 24 hours after surgery from postoperative in post anaesthesia care unit and in orthopaedic wards as primary outcome of the study.

SECONDARY OUTCOMES:
The aim of this study is to compare IPACK Block with Adductor Canal Block versus Adductor Canal Block Alone on Functional Recovery and Inflammatory Response and range of motion postoperatively | Postoperative Pain scores at rest and during active flexion 45◦ will be recorded at 8 hours, 12 hours and 24 hours postoperative.
  Assessment of pain ( by 11 point numeric pain rating scale) after completing the surgical procedure and wear off of spinal analgesia that will be confirmed by modified Bromage scale and cold sensation. Assessment of pain scores at rest and during active flexion 45◦ will be recorded at 8 hours, 12 hours and 24 hours postoperatively, patients will be asked to rate perceived pain using an 11-point Numeric Pain Rating Scale (NRS: 0= no pain and 10= worst pain) experienced at rest and during active flexion 45◦.
The aim of this study is to compare IPACK Block with Adductor Canal Block versus Adductor Canal Block Alone on Functional Recovery and Inflammatory Response and range of motion postoperatively | Range of motion and quadriceps strength will be measured after first 10 hours, three times a day with 6 hours apart.
  Range of motion and quadriceps strength (by extent of knee extension) will be measured to grade the functional recovery of the knee joint after surgery after the first 10 hours postoperatively. The extent of knee extension will be used to quantify the range of motion (ROM). The interval of activities will be recorded three times a day with 6 hours apart.
The aim of this study is to compare IPACK Block with Adductor Canal Block versus Adductor Canal Block Alone on Functional Recovery and Inflammatory Response and range of motion postoperatively. | Neutrophil-lymphocytic ratio and Platelet-lymphocytic ratio will be collected at 12 hours and 24 hours postoperative.
  Blood samples for neutrophil-lymphocytic ratio (NLR) (normal range in normal male and female are 0.43 - 2.75 and 0.37 - 2.87 respectively) and platelet-lymphocytic ratio (PLR) (normal range in male and female are 36.63 - 149.13 and 43.36 - 172.68 respectively) will be collected at 12 hours and 24 hours postoperative.

IPD SHARING:
Plan to Share IPD: Undecided